CLINICAL TRIAL: NCT04689035
Title: A Phase 1, Randomised, Double-blind, Placebo-controlled, Single Ascending Dose Study in Healthy Volunteers to Evaluate the Safety, Tolerability and Pharmacokinetics of Intravenously Administered AVLX-144
Brief Title: A Phase 1 Study in Healthy Volunteers to Evaluate the Safety, Tolerability and Pharmacokinetics of AVLX-144
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avilex Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AVLX-144CS01
Record Dates: First submitted 2020-12-15; First posted 2020-12-30 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2020-07

CONDITIONS: Safety Issues; Tolerance
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): AVLX-144_dose1
  Interventions: Drug: AVLX-144; Drug: Placebo
- Cohort 2 (Experimental): AVLX-144_dose2
  Interventions: Drug: AVLX-144; Drug: Placebo
- Cohort 3 (Experimental): AVLX-144_dose3
  Interventions: Drug: AVLX-144; Drug: Placebo
- Cohort 4 (Experimental): AVLX-144_dose4
  Interventions: Drug: AVLX-144; Drug: Placebo
- Cohort 5 (Experimental): AVLX-144_dose5
  Interventions: Drug: AVLX-144; Drug: Placebo
- Cohort 6 (Experimental): AVLX-144_elderly
  Interventions: Drug: AVLX-144; Drug: Placebo

INTERVENTIONS:
Drug: AVLX-144 — Test drug
  Other Names: Test drug
Drug: Placebo — Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled, single ascending dose study in healthy volunteer subjects. Each dose level will be investigated with eight 20-50-year-old male subjects (6 on active drug and 2 on placebo). Additionally, eight healthy elderly subjects (65-80 years of age, males and females), 6 on active drug and 2 on placebo, will be included in the study at one dose level, once the safety and tolerability of AVLX-144 has been documented in younger subjects.

ELIGIBILITY:
Inclusion Criteria:

- Healthy male and female subjects, body mass index (BMI) 18-28 kg/m2, body weight from 50 kg (females) or 60 kg (males) up to 100 kg, good general health.

Exclusion Criteria:

- History or evidence of current clinically significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, haematological, metabolic-endocrine, neurological, urogenital or psychiatric disorder. Febrile convulsions in childhood do not necessarily exclude a subject, but subjects with any type of generalized seizure in adulthood must be excluded. Personal or first-degree family history of congenital long QT syndrome or sudden death of a first-degree relative suspected to be due to long QT syndrome will also exclude the subject.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AVLX-144 | From randomisation to end of study participation
  Safety and tolerability will be assessed by recording adverse events (AEs), by performing physical examinations and safety laboratory assessments (blood and urine), and by recording vital signs and electrocardiograms (ECGs).

SECONDARY OUTCOMES:
Pharmacokinetics parameter | From dosing until 48 hours after dosing
  AUClast (the area under the plasma concentration-time curve from time zero to the last sample with a quantifiable concentration)
Pharmacokinetics parameter | 24 hrs
  AUC0-24 (the area under the plasma concentration-time curve from time zero to 24 h),
Pharmacokinetics parameter AUC | From start to end of assessment
  AUCinf (the area under the plasma concentration-time curve from time zero extrapolated to infinity, if feasible)
Pharmacokinetics parameter elimination | From start to end of assessment
  elimination constant λz and t½ (terminal elimination half-life, if feasible), and systemic plasma clearance (Cl) and volume of distribution (Vd)

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, MD, Principal Investigator — Clinical Research Services Turku - CRST Oy
Locations (1):
- Clinical Research Services Turku / CRST Oy, Turku, Finland

IPD SHARING:
Plan to Share IPD: No